CLINICAL TRIAL: NCT03249493
Title: Monitoring Of Viral Load In Decentralised Area in Vietnam : Improving Access to Viral Load Monitoring in HIV-infected Patients on ART
Brief Title: Monitoring Of Viral Load In Decentralised Area in Vietnam
Acronym: MOVIDA-2
Status: Completed | Type: Observational
Sponsor: Institut Pasteur (Industry)
Collaborators: Global Fund (Other); National Institute of Hygiene and Epidemiology, Vietnam (Other); Hanoi University of Public Health (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2016-001
Record Dates: First submitted 2017-08-07; First posted 2017-08-15 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2021-03

CONDITIONS: HIV/AIDS; Dried Blood Spot; Viral Load
Keywords: Decentralised Area
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples on Dried Blood spot cards
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HIV Injection drug users: Blood sample on DBS. Blood sample for HIV Viral Load measurements and HIV Drug Resistance at baseline, 6, 12 and 24 months of follow up after ART initiation using Dried Blood Spot
  Interventions: Other: Blood sample on DBS
- HIV Non injection drug users: Blood sample on DBS. Blood sample for HIV Viral Load measurements and HIV Drug Resistance at baseline, 6, 12 and 24 months of follow up after ART initiation using Dried Blood Spot
  Interventions: Other: Blood sample on DBS

INTERVENTIONS:
Other: Blood sample on DBS — We will take 5 mL of whole blood at ART initiation, 6, 12 and 24 months of follow up after ART initiation. Blood will be transferred on DBS cards.
  HIV Viral Load measurements will be done and HIV Drug Resistance measurements will be performed in case of 2 consecutive VL results > 1000 cp/mL

SUMMARY:
As of today, HIV-infected patients followed in decentralized area have little or even no access to viral load monitoring because laboratories able to perform this biological measurement are only in large cities, and because plasma transfer to these laboratories is complex and very costly.

Blood sampling using dried blood spots (DBS) could overcome these difficulties. The goal of this operational research is to document the feasibility of DBS use in decentralised area to monitor viral load, to evaluate the virological response on ART, and to compare the virological response between injecting drug users (IDU) and the other patients, as IDU represent a large proportion of HIV-infected patients who may have a lower access/adherence to care.

DETAILED DESCRIPTION:
The MOVIDA project is a longitudinal observational study enrolling patients who initiate ART in decentralized areas requiring individual data and blood samples collected in routine HIV care.

This project aims at evaluating and providing operability data of the use of Dried Blood Spots (DBS) as sampling tool to measure and monitor the HIV viral load in real life in rural decentralized areas in Vietnam.

This operational project would contribute to:

* the provision of viral load measurements in patients from rural decentralized areas,
* the improvement of the proportion of patients in virological success on ART, and hence to reduce the proportion of patients with acquired HIV drug resistance,
* the improvement of general HIV care and to establish an observatory of HIV drug resistance,
* strengthen national capacities through capitalization and exchange of good practices of blood sampling using DBS system to expand to other indications than HIV VL measurement.

To achieve this goal, clinical and laboratory staff will be trained to the management of the MOVIDA project (enrollment of patients; sample collection, management and analysis; data collection) before the operational observational study. Patients on the antiretroviral (ART) initiation visit will be informed about the study and invited to participate, before collection of blood to prepare DBS and collection of clinical data already routinely collected in the patient medical records. The blood collection (5ml) will be repeated at 6, 12 and 24 months during follow-up visits already planned according to the current national guidelines for the ART delivery.

The samples collected (5ml of blood) will be analyzed in a local central laboratory using the m2000rt Abbott techniques. Analysis results (VL and when necessary HIV Drug Resistance genotyping) will be available to the medical doctor in order to adapt the patient treatment appropriately. A set of randomly selected DBS will be shipped to France for centralized quality control analyses.

A socio-anthropological qualitative study will also be implemented targeting patients, health-care staff and peer health workers to apprehend their understanding of VL, and to better define determinants of adherence and attendance to clinical visits. This will help local health authorities adapt the messages and the initiatives to improve adherence to ART and attendance to care follow-up.

The study duration is 36 months with a 6 months period of enrollment and will be conducted in 6 provinces where 1000 patients are to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* confirmed HIV-1 infection,
* age at enrolment ≥18 years,
* ART naïve (women exposed through PMTCT are eligible),
* consent to participate.

Exclusion Criteria:

* negative for HIV,
* age at enrolment <18 years,
* ART experienced (excepted PMTCT),
* not consenting to participate.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The key population for this research project is HIV-positive patients who initiate ART followed in 24 out-patient clinics (OPCs) located in decentralised areas in two provinces, where laboratories facilities are not easily accessible and where VL monitoring is extremely scarce.
Sampling Method: Non-Probability Sample
Enrollment: 584 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Virological success at 24 months of ART | 24 months (+/- 1 month) after ART initiation
  Patients with a VL <1000 copies/mL at 24 months of ART

SECONDARY OUTCOMES:
Outcomes related to DBS transfer | through study completion, an average of 2 years
  * Delay (days) between DBS collection and transfer to central laboratory
  * Delay (days) between DBS collection and reception at central laboratory
Outcomes related to quality of DBS samples | through study completion, an average of 2 years
  - Aspect of DBS at reception at central laboratory (qualitative evaluation)
Outcomes related to delay concerning the return of viral load result | through study completion, an average of 2 years
  * Delay (days) between reception at central laboratory and viral load quantification
  * Delay (days) between DBS collection and reception of the result at the care site
Outcomes related to ability of DBS to provide viral load result | through study completion, an average of 2 years
  - Proportion of DBS not allowing viral load quantification (number of DBS not allowing VL quantification/total number of DBS samples)
Outcomes related to ability of DBS to provide HIV drug resistance result | through study completion, an average of 2 years
  - Proportion of DBS not allowing HIV drug resistance (number of DBS not allowing HIV drug resistance /total number of DBS samples with VL confirmed>1000cp/mL)
Impact of viral load result on second-line ART initiation | through study completion, an average of 2 years
  - Number of patients who initiate second-line ART during the study
Impact of viral load result on second-line ART initiation in term of delay | through study completion, an average of 2 years
  - Delay (days) between reception of the viral load results at the care site and second-line ART initiation
virological success at 6 and at 12 months of ART | At 6 and 12 months of ART
  Patients with a VL <1000 copies/mL at 6 and at 12 months of ART
Virological failure at 6, 12 and 24 months of ART | At 6, 12 and 24 months of ART
  - Proportion of patients with 2 consecutive viral load >= 1000 copies/mL (the second viral load being measured within 2 to 3 months from the first one after strengthening of adherence)
HIV drug resistance in case of virological failure at 6, 12 and 24 months of ART | At 6, 12 and 24 months of ART
  - Proportion of patients in virological failure and for whom the virus is harbouring HIV drug resistances
Description of HIV drug resistance in case of virological failure at 6, 12 and 24 months of ART | At 6, 12 and 24 months of ART
  - Profiles of HIV durg resistance in patients in virological failure
Baseline HIV drug resistance in case of virological failure | ART initiation
  - Proportion of patients identified in virological failure during the follow-up on ART, and for whom the virus presented HIV drug resistance at ART initiation
Baseline HIV drug resistance | ART initiation
  - proportion of patients for whom the virus presented HIV drug resistance at ART initiation, in a random selection of patients enrolled
Mortality | through study completion, an average of 2 years
  Patients who died while on ART during the follow-up
Attrition | through study completion, an average of 2 years
  patients who are lost to follow-up (not seen for >3 months) after they initiated ART

CONTACTS AND LOCATIONS:
Overall Officials: Fabien TAIEB, MD, Principal Investigator — Institut Pasteur; Yoann Madec, PhD, Principal Investigator — Institut Pasteur
Locations (1):
- Yen Bai medical center, Yên Bái, Vietnam

IPD SHARING:
Plan to Share IPD: No
Non applicable

REFERENCES:
- [Background] Taieb F, Tran Hong T, Ho HT, Nguyen Thanh B, Pham Phuong T, Viet Ta D, Le Thi Hong N, Ba Pham H, Nguyen LTH, Nguyen HT, Nguyen TT, Tuaillon E, Delaporte E, Le Thi H, Tran Thi Bich H, Nguyen TA, Madec Y. First field evaluation of the optimized CE marked Abbott protocol for HIV RNA testing on dried blood spot in a routine clinical setting in Vietnam. PLoS One. 2018 Feb 9;13(2):e0191920. doi: 10.1371/journal.pone.0191920. eCollection 2018. PMID 29425216
- [Background] Taieb F, Tram TH, Ho HT, Pham VA, Nguyen L, Pham BH, Tong LA, Tuaillon E, Delaporte E, Nguyen AT, Bui DD, Do N, Madec Y. Evaluation of Two Techniques for Viral Load Monitoring Using Dried Blood Spot in Routine Practice in Vietnam (French National Agency for AIDS and Hepatitis Research 12338). Open Forum Infect Dis. 2016 Jul 7;3(3):ofw142. doi: 10.1093/ofid/ofw142. eCollection 2016 Sep. PMID 27704001
- [Result] Nguyen TA, Tran TH, Nguyen BT, Pham TTP, Hong Le NT, Ta DV, Phan HTT, Nguyen LH, Ait-Ahmed M, Ho HT, Taieb F, Madec Y; MOVIDA 2 study group. Feasibility of dried blood spots for HIV viral load monitoring in decentralized area in North Vietnam in a test-and-treat era, the MOVIDA project. PLoS One. 2020 Apr 9;15(4):e0230968. doi: 10.1371/journal.pone.0230968. eCollection 2020. PMID 32271796
- [Derived] Araujo Chaveron L, Pham TTP, Nguyen BT, Tran TH, Le NTH, Pham TH, Ngo KP, Tong HT, Phan HTT, Ait-Ahmed M, Nguyen TA, Taieb F, Madec Y; MOVIDA 2 study group. Injecting drug use increases the risk of death in HIV patients on antiretroviral therapy in Vietnam. AIDS Care. 2024 May;36(5):631-640. doi: 10.1080/09540121.2023.2224549. Epub 2023 Jun 20. PMID 37339000
- [Derived] Lefrancois LH, Nguyen BT, Pham TTP, Le NTH, Dao HTT, Tran TH, Ngo KP, Tong HT, Phan HTT, Ait-Ahmed M, Pham TH, Nguyen TA, Taieb F, Madec Y; MOVIDA 2 study group. Assessment of HIV viral load monitoring in remote settings in Vietnam - comparing people who inject drugs to the other patients. PLoS One. 2023 Feb 21;18(2):e0281857. doi: 10.1371/journal.pone.0281857. eCollection 2023. PMID 36802388